CLINICAL TRIAL: NCT06147362
Title: 68Ga-NOTA-PEG2-RM26 PET/CT: Tracer Biodistribution and Uptake in Different Kinds of Cancer With Gastrin-Releasing Peptide Receptor (GRPR) Overexpression
Brief Title: 68Ga-NOTA-PEG2-RM26 PET/CT, First in Man Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Stockholm South General Hospital (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Jeffrey Yachnin M.D., PhD., Section Head Early Clinical Trial Unit, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2021-004980-28
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Approximately ten patients (with primary/recurrent or metastatic cancer) in each of the following six cancer groups, prostate cancer, breast cancer, colorectal cancer, gastrointestinal carcinoid, gastric cancer, and lung cancer, will be recruited and examined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-PEG2-RM26 (Experimental): Participants will be injected with 2 MBq/kg of 68Ga-NOTA-PEG2-RM26 limited to 100-200 MBq and then undergo PET/CT examination.
  Interventions: Drug: 68Ga-NOTA-PEG2-RM26

INTERVENTIONS:
Drug: 68Ga-NOTA-PEG2-RM26 — Single-dose 68Ga-NOTA-PEG2-RM26, a gastrin-releasing peptide receptor antagonist linked with a positron emitting radioisotope intravenously injected into participants before the PET/CT scans.

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-PEG2-RM26 in prostate cancer patients. A single dose of 2 MBq/kg of 68Ga-NOTA-PEG2-RM26 limited to 100-200 MBq per examination will be given intravenously. Visual and semiquantitative method will be used to assess PET/CT images.

DETAILED DESCRIPTION:
The gastrin-releasing peptide receptor (GRPR), also known as bombesin receptor subtype II (BB2), is a member of the G protein-coupled receptor family of bombesin receptors. GRPR is over-expressed in various types of human tumors. RM26, a GRPR antagonist with high affinity, was discovered by peptide backbone modification of bombesin analogues.

To target gastrin-releasing peptide receptor in human neoplastic cells NOTA-PEG2-RM26 was synthesised and then labeled with 68Ga.

An open-label whole-body PET/ CT study was designed to investigate the safety and dosimetry of 68Ga-NOTA-PEG2-RM26 and to assess its clinical diagnostic value in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Primary/recurrent or metastatic cancer in: prostate cancer, breast cancer, colorectal cancer, gastrointestinal carcinoid, gastric cancer, or lung cancer
* Histopathological diagnosis
* Age 18 years or more and palliative disease OR age above 50 years
* Adequate bone marrow, hepatic and renal function, Eastern Cooperative Oncology Group Performance Status Scale 0 or 1 and a negative pregnancy test

Exclusion Criteria:

* Age less than 18 years
* Less than 6 months since a clinically significant cardiovascular event such as myocardial infarction, unstable angina, angioplasty, bypass surgery, stroke or transient ischemic attack
* Congestive heart failure New York Heart Association class ≥ II
* Pregnant or breast-feeding women
* Patients with reproductive potential not implementing accepted and effective means of contraception
* Participation in any other clinical trial within the previous 4 weeks
* Unable to comply with study procedures (e.g., claustrophobia, low back pain not allowing the patient to lay down in the examination bed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events within 2 weeks of injection | 2 weeks
  Adverse events within 2 weeks of injection and scanning of participants

SECONDARY OUTCOMES:
Biodistribution of 68Ga-NOTA-PEG2-RM26 | During procedure
  The semiquantitative analysis will be performed by the same person for all the cases, uptake in organs with uptake above the blood pool will bes described
Dosimetry of 68Ga-NOTA-PEG2-RM26 | During procedure
  Mean absorbed radiation doses will be estimated using the source and target organ framework outlined by the Medical Internal Radiation Dose Committee. Absorbed and effective radiation doses will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yachnin, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided